CLINICAL TRIAL: NCT05335018
Title: Phase II Study of Glofitamab, Poseltinib and Lenalidomide in Patients with Relapsed/refractory Diffuse Large B Cell Lymphoma
Brief Title: GPL in Patients with Relapsed/refractory Diffuse Large B Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sung-Soo Yoon, hematology oncology Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPL
Record Dates: First submitted 2022-03-24; First posted 2022-04-19 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Relapsed/refractory Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — glofitamab; poseltinib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): total 2years. Glofitamab: Increase from 2.5mg for 8days in 1 cycle to 10mg for 15days. 2cycles 1day 30mg, 30 mg on the 1st day of every week thereafter. Poseltinib: 40mg/day bid orally, administered daily from the 1st to the 21st of every week.
  Lenalidomide: 20mg/day bid orally, administered daily from the 1st to the 14st of every week.
  Interventions: Drug: Glofitamab, Poseltinib, Lenalidomide

INTERVENTIONS:
Drug: Glofitamab, Poseltinib, Lenalidomide — Glofitamab: Increase from 2.5mg for 8days in 1 cycle to 10mg for 15days. 2cycles 1day 30mg, 30 mg on the 1st day of every week thereafter. Poseltinib: 40mg/day bid orally, administered daily from the 1st to the 21st of every week.
  Lenalidomide: 20mg/day bid orally, administered daily from the 1st to the 14st of every week.

SUMMARY:
Prospective, open-ended, single-arm, multicenter Phase II clinical trial. To evaluate the efficacy of Glofitamab, Poseltinib, and Lenalidomide combination therapy in patients with relapsed/refractory diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
For outpatients or inpatients who meet the criteria for subject selection, the study is conducted with patients who have given a sufficient explanation of the study and who voluntarily consented to participate in the study.

Patients enrolled in the study receive a combination therapy of glofitamab, poseltinib, and lenalidomide according to the criteria specified in the protocol.

This therapy is defined as one cycle of 3 weeks, and a total of 12 cycles is planned.

glofitamab is administered in steps. 2.5 mg on the 8th day of Cycle 1, 10 mg on the 15th day, 30 mg on the 1st day of Cycle 2, and then 30 mg intravenously on the 1st day of each cycle.

poseltinib is administered orally at 40 mg BID daily from Day 1 to Day 21 of each cycle, and lenalidomide is administered orally at 30 mg QD daily from Day 1 to Day 14 of each cycle.

Maintenance therapy is offered with poseltinib and lenalidomide only for patients with a partial response (PR) or complete response (CR).

In addition, this study includes a salvage protocol for patients with CNS (central nerve system) lesions during patient recruitment.

These patients are excluded from treatment with glofitamab because of the potential risk of CNS toxicity and will receive only poseltinib plus lenalidomide.

The first 3+3 patients will proceed to a safety cohort, with dose adjustments for lenalidomide and poseltinib. These 6 persons were not included in the cohort evaluating the outcome of the study.

ELIGIBILITY:
1. Inclusion Criteria

   * Male and female aged ≥19 years

     * Histologically diagnosed with CD20-expressing B-cell NHL

       -Diffuse large B-cell lymphoma (DLBCL)
       * Transformed follicular lymphoma

         * Relapse after or failure to respond to at least prior treatment regimen treatments and last dose administered must be more than 2-weeks ahead from enrollment
       * Should have received anti-CD20 based chemotherapy previously
       * Failed to at least two lines of therapy if patient is candidate for autologous stem cell transplantation
       * Failed frontline therapy if patient is ineligible for autologous stem cell transplantation.

         ④Not eligible if patient's IHC expression is both BCL6(-) and MYC(+). However, in the salvage cohort group, subjects with previous pathological test results of BCL6(-) and MYC(+) may be eligible.

         ⑤Measurable disease, defined as at least one bi-dimensionally measurable nodal lesion, defined as > 1.5 cm in its longest dimension, or at least one bi-dimensionally measurable extranodal lesion, defined as > 1.0 cm in its longest dimension.

         ⑥Eastern Cooperative Oncology Group (ECOG) status of 0, 1, or 2

         ⑦Adequate liver, hematological and renal function.
       * Total bilirubin ≤ 2 x ULN and AST, ALT ≤ 3 x ULN
       * WBC ≥ 3,000 /μL, ANC ≥ 1,000 /μL, Platelets ≥ 75,000 /μL, and Hemoglobin ≥ 9.0 g/dL. (adjustment with blood transfusion & G-CSF within 2 weeks is not allowed)
       * Cr ≤ 1.5 x ULN or CLcr ≥ 30 mL/min (Cockcroft-Gault)

         * Negative test results for Hepatitis C virus (HCV) antibody. ⑨Negative test results for human immunodeficiency virus (HIV).

           * Sexually active women of childbearing potential (WOCPB) should have 2 negative urine hCG tests before administration of the study intervention. Tests should be conducted every week for the first month of the study, then every 4 weeks thereafter, or every two weeks in case of irregular menstruation. Urine hCG tests should be performed through 4 weeks after the last dose of glofitamab, poseltinib, or lenalidomide, whichever comes later. WOCPB should use 2 contraceptive methods, including at least 1 highly effective contraceptive method, for 4 weeks before the first dose, during the treatment period, 4 weeks after the last dose of poseltinib and lenalidomide, 2 months after the last dose of glofitamab, and 18 months after the last dose of obinutuzumab. Women who is menopause (no menstruation for at least 12 months, not related to drug) or surgically sterile (have no ovaries or no uterus or neither) are not required to undergo pregnancy tests. Sexually active men should use condoms during the treatment period and until 4 weeks after the last dose of poseltinib and lenalidomide, 2 months after the last dose of glofitamab, and 3 months after the last dose of obinutuzumab.

             ⑪Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules.
             * Is able to understand the purpose and risks of the study and to authorize the use of his/her medical information for the purpose of the study.
2. Exclusion Criteria

<!-- -->

1. Has previously received 4 or more lines of anticancer chemotherapies (autologous hematopoietic stem cell transplantation is considered as 1 line of treatment).
2. Has current evidence or history of macrophage activation syndrome/hemophagocytic lymphohistiocytosis (MAS/HLH).
3. Prior treatment with glofitamab.
4. Has acute bacterial, viral, or fungal infections confirmed with positive blood culture or diagnosed clinically in case there is no positive blood culture.
5. Has known active infection or reactivation of latent infection, regardless of bacteria, viruses, fungi, mycobacteria, or other pathogens, or has an episode of major infection requiring hospitalization or intravenous antibiotic treatment within 4 weeks from the dose of study drug.
6. Has received systemic immunotherapy including a radioimmunoconjugate, an antibody-drug conjugate, or an immune checkpoint inhibitor (eg. anti-cytotoxic T-lymphocyte-associated protein 4 [anti-CTLA4], anti-programmed death 1 [anti-PD1], and anti-programmed death ligand 1 [anti-PDL1]) within 4 weeks from the dose of study drug or within 5 half-lives of the drug.
7. Has experienced treatment-emergent immune-related AE during previous immunotherapy.
8. Has received radiotherapy, anticancer chemotherapy, or other experimental chemotherapy including chimeric antigen receptor therapy (CAR-T) within 4 weeks from the first dose of study drug.
9. Has received a homologous hematopoietic stem cell transplantation within 1 year or has previously received a solid organ transplantation.
10. Has received autologous hematopoietic stem cell transplantation within 100 days from the first dose of study drug.
11. Has a graft-versus-host disease (GVHD) requiring treatment.
12. Is not able to have oral intake of study drug.
13. Has resistance to BTK inhibitors or lenalidomide (defined as PFS less than 6 months after BTK inhibitors or lenalidomide).
14. Has previously been diagnosed with a malignancy other than the cancer included in this study, except appropriately treated basal cell carcinoma, squamous cell skin cancer, in situ cancer, and at least 5 years of disease free status from previous cancer.
15. Has a clinically significant cardiovascular disease as follows: a heart disease of New York Heart Association Functional Class III or IV or Objective class C or D, or had myocardial infarction within 6 months, or has uncontrolled arrhythmia or unstable angina. Of note, patients with well-controlled and asymptomatic atrial fibrillation are eligible.
16. Malabsorption syndrome, diseases that seriously affect gastrointestinal function, resection of the stomach or small intestine that may affect absorption, inflammatory bowel disease with symptoms, partial or complete intestinal obstruction, or obesity surgery such as gastric restriction and gastric bypass surgery.
17. Has a history of drug-specific hypersensitivity or anaphylaxis to the study drug (including active ingredients or excipients).
18. A condition with uncontrolled active bleeding or potential bleeding (e.g., hemophilia or von Willebrand disease)
19. Uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP).
20. Requiring treatment with a strong cytochrome P450 (CYP)3A4 inhibitor/inducer.
21. Is receiving or needs to receive warfarin or a corresponding vitamin K antagonist (e.g., phenprocoumon within 7 days from the first dose of study drug.
22. Prothrombin time (PT)/international normalized ratio (INR) or activated partial thromboplastin time) (aPTT) (in the absence of lupus anticoagulant) >2x ULN
23. Needs to receive a proton pump inhibitor (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole).Patients receiving proton pump inhibitors will be eligible after changing regiment to H2-receptor antagonists or antacids.
24. History of cerebrovascular disease or event including stroke or intracranial hemorrhage within 6 months prior to the first dose of study drug.
25. Has underwent major surgery within 28 days of the first dose of study drug. Subjects who underwent major surgery should be properly recovered prior to the first dose of the drug.
26. Serological status of hepatitis B or hepatitis C: If HBsAg is positive, the subject may be enrolled if he/she is on appropriate antiviral treatment and HBV DNA is not detectable. Patients who are HBcAb-positive, HBsAg-negative, and HBV DNA-negative should receive appropriate antiviral preventive treatment during the study. Patients who are positive for hepatitis C antibodies should have negative PCR results, and those with positive PCR results will be excluded. However, the salvage cohort group does not require preventive treatment. For safety, patients will continue active anti-HBV treatment with HBV DNA tests performed every 3 months until at least 6 months after completion of hie/her study participation. HBV DNA will be tested by PCR.
27. Has an active tuberculosis (a history of exposure or a history of positive tuberculosis testing with clinical symptoms or physical or radiological findings) or a latent tuberculosis requiring treatment.
28. Has a primary or secondary CNS lymphoma at enrollment.
29. Has active or a history of CNS disease with stroke, epilepsy, CNS vasculitis, or neurodegenerative disease. Patients with a history of stroke will be eligible if he/she has been without a stroke or transient ischemic attack in the past 2 years and no neurological deficits. However, patients with CNS involvement but there is no relevant CNS disease or patients who have not experienced related symptoms may be eligible. In addition, if there is CNS involvement, but registration in the main cohort is possible, registration in the main cohort can be done after discussion with the state responsible agency. In addition, patients with CNS involvement but there is possible to register in the main cohort, it can be registered in the main cohort after discussion with the investigator of mainstudy site.
30. Has a significant and uncontrolled disease that may affect compliance with the study protocol or interpretation of the results, including diabetes, lung disease, and autoimmune diseases.
31. Has received attenuated live vaccine within 4 weeks prior to the first dose of study drug, or is expected to require attenuated live vaccine during the study.
32. Has received systemic immunosuppressive drugs (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to the first dose of study drug. Prednisone ≤ 25 mg/day or equivalent corticosteroid treatment is allowed.
33. Has a history of autoimmune disease, including but not limited to myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with a medical history of distant past autoimmune diseases or a current well-controlled autoimmune disease may be enrolled after discussing and checking with the Monitor.
34. Has diseases in which the use of the study drug is contraindicated or other illness, metabolic disorders, physical examination findings, or clinical examination findings with suspected such conditions.
35. Is breastfeeding or pregnant.
36. Is participating in another therapeutic clinical trials.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy evaluation of Gofitamab, Poseltinib, and Lenalidomide using endpoints | At the end of Cycle 2 (each cycle is 28 days)
  Overall Response Rate according to Lugano criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sung-soo Yoon, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea